CLINICAL TRIAL: NCT04643782
Title: A Single Arm, Open-Label, Multi-Center, and Comparative Study of the Anne Sleep System Versus Polysomnography to Diagnose Obstructive Sleep Apnea: ANNE Program for the Non-Invasive Evaluation of Apnea in Sleep (APNEAs)
Brief Title: Comparative Study of the ANNE™ One System to Diagnose Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Sibel Health Inc. (Industry)
Responsible Party: Principal Investigator, Phyllis Zee, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU0021444
Record Dates: First submitted 2020-11-16; First posted 2020-11-25 (Actual); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Intervention Model Description: Patients will use ANNE Sleep system during one night of polysomnography recording in sleep lab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm Study (Other): After consent, subjects will wear the ANNE sleep system during an attended PSG study for 1 night.
  Interventions: Device: ANNE Sleep

INTERVENTIONS:
Device: ANNE Sleep — ANNE sleep system

SUMMARY:
The main objective of this study is to evaluate the accuracy of the ANNE Sleep system for the diagnosis of obstructive sleep apnea (OSA) in adults

DETAILED DESCRIPTION:
The main object of this study is to evaluate the accuracy of the ANNE Sleep system for the diagnosis of obstructive sleep apnea (OSA) in adults. Our primary hypothesis is that the ANNE Sleep system is non-inferior compared to polysomnography (PSG) for the diagnosis of obstructive sleep apnea

ELIGIBILITY:
Inclusion Criteria:

1. ≥22 years old.
2. Subjects with suspected OSA based on history and physical who qualify for, and have either a PSG or HSAT ordered, as determined by their regular provider. Subjects with self-reported symptoms of OSA based on the STOP-Bang questionnaire indicating affirmative answers to any of the following: snoring, daytime fatigue/sleepiness/tiredness, partners who have observed the subject stopping breathing or choking/gasping during sleep. Persons with a previous diagnosis of OSA are also eligible.
3. Willingness to give written consent and comply with study procedures

Exclusion Criteria:

1. An unstable medical condition, acute or chronic, that in the opinion of the investigator puts the subject at health risks related to this trial or interferes with the clinical trial and data collection
2. Inability to understand instructions
3. Has a skin abnormality that precludes assessment
4. Has a history of dementia
5. Patients with implanted pacemakers or defibrillators
6. Subject is pregnant, nursing or planning a pregnancy over the expected course of the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois
  - Carle Foundation Hosipital, Urbana, Illinois
  - Central Dupage Hospital (CDH), Winfield, Illinois

IPD SHARING:
Plan to Share IPD: No
Data stored and used for future research will be de-identified. Data will not be used for future research outside of the scope of this study.

REFERENCES:
- [Derived] Davies C, Lee JY, Walter J, Kim D, Yu L, Park J, Blake S, Kalluri L, Cziraky M, Stanek E, Miller J, Harty BJ, Schauer J, Rangel SM, Serao A, Edel C, Ran DS, Olagbenro MO, Lim A, Gill K, Cooksey J, Toloui O, Power T, Xu S, Zee P. A single-arm, open-label, multicenter, and comparative study of the ANNE sleep system vs polysomnography to diagnose obstructive sleep apnea. J Clin Sleep Med. 2022 Dec 1;18(12):2703-2712. doi: 10.5664/jcsm.10194. PMID 35934926

RESULTS

PARTICIPANT FLOW:
Groups:
- ANNE Sleep System: After consent, subjects will wear the ANNE sleep system during an attended PSG study for 1 night.
  ANNE Sleep: ANNE sleep system
Period: Overall Study
Arm/Group | ANNE Sleep System
Started | 287
Completed | 225
Not Completed | 62

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 202
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 26
  White | 164
  More than one race | 10
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 225

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Obstructive Sleep Apnea (OSA) Diagnosis Using ANNE Sleep System Compared to Polysomnography
Description: The diagnosis of moderate to severe OSA by determining a patient's Apnea-Hypopnea Index (AHI) using the ANNE Sleep system compared to Polysomnography (PSG) over one (1) night worn concurrently.
  Sensitivity is the number of true positives divided by the sum of the number of true positives and false negatives. Specificity is the number of true negatives divided by the sum of the number of true negatives and false positives.
Time Frame: 1 night
Measure: Mean (95% Confidence Interval); unit: percentage of true cases
Arm/Group | Single Arm Study
Number analyzed (Participants) | 225
percentage of true cases
  Sensitivity | 89.7 [79.9 to 95.8]
  Specificity | 97.5 [93.6 to 99.3]

ADVERSE EVENTS:
Time Frame: One night of sleep.
Description: Subjects wear the ANNE Sleep device concurrently with the gold standard polysomnography over one night of sleep.
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/225
Serious Adverse Events (participants affected / at risk) | 0/225
Other Adverse Events (participants affected / at risk) | 0/225

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04643782/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04643782/ICF_001.pdf